CLINICAL TRIAL: NCT00785369
Title: In Vivo Reflectance Confocal Microscopy for Pigmented Lesion Diagnosis: A Multi-center Study
Brief Title: In Vivo Confocal Microscopy for Pigmented Lesion Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucid, Inc. (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Loma Linda University (Other); University of Rochester (Other); VA Loma Linda Health Care System (U.S. Federal Agency); Skin and Cancer Associates in Plantation,Fl. (Unknown); Harvard University (Other)
Responsible Party: Sponsor
Organization: Lucid (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LI058054; 5R44CA058054-06 (NIH)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Skin Cancer; Melanoma; Lentigo Maligna
Keywords: skin disorders; skin cancer; melanoma; lentigo maligna
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Hutchinson's Melanotic Freckle; Skin Diseases | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Device: In vivo reflectance confocal microscopy of pigmented lesions in vivo
  Interventions: Device: Reflectance confocal microscopy

INTERVENTIONS:
Device: Reflectance confocal microscopy — Reflectance confocal microscopy (VivaScope 1500)
  Other Names: Device

SUMMARY:
The purpose of this study is to image pigmented skin lesions suspicious for melanoma with an imaging technology called in vivo reflectance confocal microscopy. This technology uses low intensity laser to image below the surface of the skin. The confocal images of the suspicious skin lesion will be examined. The goal of this study is to compare the results of the confocal image examination to the pathologic diagnosis of the skin lesion.

The technique being evaluated in this study uses reflectance confocal microscopy in vivo. The term "in vivo" means in/on a living subject. In this study you will be the living subject and the confocal microscope will be placed on your skin to look at your skin lesion. The confocal microscope uses a weak laser light and a sophisticated lens to image the individual cells that make up the skin. Your lesion will be photographed with high resolution photography.

DETAILED DESCRIPTION:
Patients will be imaged with the VivaScope 1500 reflectance confocal microscope during a single patient visit. The lesion will be photographed with high resolution photography and a high resolution dermoscopic device.

The lesion will then be prepared for RCM imaging. A skin contact device consisting of a metal ring and window will be applied to the skin surrounding the lesion of interest with a disposable medical grade adhesive. A wetting solution will be placed onto the skin. The wetting solutions include a high index oil such as a clear cosmetic oil or mineral oil. A wetting solution such as ultrasound gel will also be placed on the lens of the microscope. Application of these agents diminishes artifacts caused by light scattering at the skin surface. RCM images of the lesion will be captured through the window/contact device using the Vivascope 1500 reflectance confocal microscope provided by Lucid, Inc. Two types of images will be collected, mosaics and stacks. Mosaics are 12x12 confocal images that are optically combined or "stitched" together to create a seamless representation of a 6mm x 6mm total area at specific depths within the skin. Stacks are 0.5mm x 0.5mm confocal images taken at 5 micron intervals from the keratin layer to the superficial dermis. Mosaics and stacks will be acquired for the skin lesion. The total estimated imaging time for a patient in this study is about 10 minutes for each lesion. More than one lesion may be imaged per patient.

After the imaging is complete, the lesion will be biopsied. All lesion images will be saved on a network server for later review and analysis. All imaging will be completed by trained research staff familiar with confocal imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing biopsy for a pigmented lesion suspicious for malignancy.
* Patients undergoing biopsy on an anatomical site that is readily accessible to the VivaScope 1500 (for example, chest, back, legs, arms, cheek, forehead).
* Ability to give informed consent.

Exclusion Criteria:

* Lesion suspicious for melanoma located on a site that is not amenable to confocal imaging (for example, adjacent to the nose, ears or eyes, fingers, toes).
* The lesion (suspicious for melanoma) is located on soles of the feet or palms of the hands.
* Inability to give informed consent.
* Known hypersensitivity to adhesive rings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the diagnostic accuracy of reflectance confocal scanning laser microscopy(RCM) for melanoma diagnosis when compared to the "gold standard" histopathologic diagnosis. | Once while on study

SECONDARY OUTCOMES:
To assess interobserver variability associated with interpreting confocal images for detecting cutaneous melanoma and to assess confocal correlations in a qualitative manner. | Once while on study

CONTACTS AND LOCATIONS:
Overall Officials: Allan C Halpern, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Center, Manhattan; Ashfaq Marghoob, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center, Hauppauge; Abel Torres, MD, Principal Investigator — Loma Linda Univeristy Adventist Health Sciences Center; Lisa Beck, MD, Principal Investigator — University of Rochester; Harold S Rabinovitz, MD, Principal Investigator — Skin and Cancer Associates, Plantation Fl.; Abel Torres, MD, Principal Investigator — VA Loma Linda Health Care System
Locations (6):
- United States (6):
  - Loma Linda University, Loma Linda, California
  - VA Loma Linda Health Care System, Loma Linda, California
  - Skin and Cancer Assoicates, Plantation, Florida
  - Memorial Sloan-Kettering Cancer Center, Hauppauge, New York
  - Memorial Sloan-Kettering Cancer Center, Manhattan, New York
  - University of Rochester Medical Center, Rochester, New York